CLINICAL TRIAL: NCT01372488
Title: Are Patients Willing and Capable of Removing Their Own Non-absorbable Sutures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fraser Health (Other)
Collaborators: University of British Columbia (Other)
Responsible Party: Principal Investigator, Peter MacDonald, Emergency Physician, Fraser Health
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2010-004
Record Dates: First submitted 2010-02-09; First posted 2011-06-14 (Estimated); Last update posted 2021-10-12 (Actual); Status verified 2021-10

CONDITIONS: Suture Removal
Keywords: Suture self removal; non-absorbable sutures
MeSH Terms: interventions — Ambulatory Care Facilities

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Study group (Active Comparator): Study group will be provided with suture removal instructions and suture removal kit and asked to consider removing their own sutures
  Interventions: Procedure: Suture self removal
- Control group (Placebo Comparator): Control group will be asked to have their sutures removed as they normally would (see family doctor or clinic)
  Interventions: Procedure: Suture removal by family doctor or clinic

INTERVENTIONS:
Procedure: Suture self removal — Suture self removal
  Arms: Study group
Procedure: Suture removal by family doctor or clinic — As above
  Arms: Control group

SUMMARY:
1. Hypothesis

   If patients who are sutured with non-absorbable sutures in the Emergency Department (ED) are provided with the proper equipment and knowledge on how to remove their own sutures, they will be willing and capable of removing their own sutures.
2. Primary and Secondary Questions

Primary Question What number of patients in the study group will successfully remove their own sutures if they are provided with the equipment and information on how to do so compared with a control group who are treated and advised in the usual fashion? (follow up with family doctor or local medical clinic for suture removal)

Secondary Questions

1. Number of complications related to self removal of sutures as compared to traditional treatment. Complications measured were wound infections, dehiscence and prolonged bleeding (>30 min)
2. Number of physician visits related to self removal of sutures as compared to traditional treatment.
3. Patient satisfaction and comfort level related to self removal of sutures as compared with traditional treatment.

DETAILED DESCRIPTION:
Introduction/Background:

Patients who are sutured with non-absorbable sutures in the Emergency Department are asked to follow up with their family doctor or local medical clinic for suture removal. Suture removal, especially for simple lacerations is easy to do. Given the proper instructions and equipment suture removal could be done by the patient or a family member.

Objectives:

Are patients willing and capable of removing their own non-absorbable sutures? How many patients can successfully self remove their own sutures if given the proper equipment and instructions as compared with patients who are not given equipment and instructions? Would patient self removal result in less physician visits related to sutured wounds? What would be the complication rate for self removal of sutures be? Specific complications were wound infection, dehiscence and prolonged bleeding? Would patients be satisfied and comfortable in taking out their own sutures?

Methods:

Patients who are sutured with non absorbable sutures in the emergency department will be randomly enrolled into either of two groups. One group will receive wound care instructions alone. The second group will be given wound care instructions, a suture removal kit and instructions regarding self-removal to take home. Both groups will be contacted by telephone 14 days after suturing and asked questions concerning who removed their sutures, number of physician visits, time loss from work related to suture removal and complications related to sutures or suture removal. Questions regarding patient satisfaction with respect to self removal of sutures will also be asked.

ELIGIBILITY:
Inclusion Criteria:

Patients 19 years and older that have wounds sutured in the ER with non-absorbable sutures

Exclusion Criteria:

* Inability to give consent secondary to alcohol, drugs or failure to speak English
* Complicated lacerations or lacerations which require close medical supervision
* Lacerations that are inaccessible to the patient (ie. scalp, back or buttock lacerations)
* Inability to contact patient by telephone for follow-up (no telephone, patient travelling out of country etc.)
* Patients who are immunocompromised, have diabetes mellitus or are on steroid medications

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2010-04; Primary Completion 2010-09 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Are patients willing and capable of removing their own non-absorbable sutures? | 3 months
  What number of patients in the study group will successfully remove their own sutures if they are provided with the equipment and information on how to do so compared with a control group who are treated and advised in the usual fashion? (follow up with family doctor or local medical clinic for suture removal)

SECONDARY OUTCOMES:
Complications related to self removal of sutures | 3 months
  Number of complications related to self removal of sutures as compared to traditional treatment were measured. Complications measured were wound infections, dehiscence and prolonged bleeding (>30 min)
Physician Visits Related to Suture Self Removal | 3 months
  Number of physician visits related to self removal of sutures as compared to traditional treatment.
Patient Comfort and Satisfaction with Self-Removal of Sutures | 3 months
  Patient satisfaction and comfort level related to self removal of sutures as compared with traditional treatment. Measures used were a survey with a 5 choice answer.

CONTACTS AND LOCATIONS:
Overall Officials: Peter J Macdonald, MD, Study Director — Royal Columbian Hospital Department of Emergency Medicine, New Westminster, BC, Canada
Locations (1):
- Royal Columbian and Eagle Ridge Hospitals, New Westminster, British Columbia, Canada

REFERENCES:
- [Result] Albert, M., Daly, A., Krueger, J., Krueger, K., Meeusen, C., Vogelheim, C., & Jones, J. (2009). 421: Self-removal of sutures by emergency department patients. Annals of Emergency Medicine, 54(3S), 133-133.